CLINICAL TRIAL: NCT00854360
Title: Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multi-Center, Dose-Range-Finding Study to Assess the Efficacy and Safety of BDP HFA Nasal Aerosol in Adult and Adolescent Patients (12 Years and Older) With Seasonal Allergic Rhinitis (SAR)
Brief Title: Study to Assess the Efficacy and Safety of BDP HFA Nasal Aerosol in Patients 12 Years and Older With SAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-AR-201
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-04

CONDITIONS: Seasonal Allergic Rhinitis; Hayfever
Keywords: Seasonal Allergic Rhinitis; Hayfever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BDP HFA 80 µg/day (Experimental): During the 2-week double-blind Treatment Period participants self-administered two actuations (one per nostril) of 40 micrograms (µg) BDP HFA and two actuations of placebo HFA once daily.
  Interventions: Drug: Beclomethasone dipropionate HFA Nasal Aerosol; Drug: Placebo
- BDP HFA 160 µg/day (Experimental): During the 2-week double-blind Treatment Period participants self-administered four actuations (two per nostril) of 40 µg BDP HFA once daily.
  Interventions: Drug: Beclomethasone dipropionate HFA Nasal Aerosol
- BDP HFA 320 µg/day (Experimental): During the 2-week double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 µg BDP HFA once daily.
  Interventions: Drug: Beclomethasone dipropionate HFA Nasal Aerosol
- Placebo (Placebo Comparator): During the 2-week double-blind Treatment Period participants self-administered four actuations (two per nostril) of placebo HFA once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beclomethasone dipropionate HFA Nasal Aerosol — Beclomethasone dipropionate (BDP) Hydrofluoroalkane (HFA) Nasal Aerosol
  Other Names: QNASL(TM)
  Arms: BDP HFA 160 µg/day; BDP HFA 320 µg/day; BDP HFA 80 µg/day
Drug: Placebo — HFA Vehicle Aerosol
  Arms: BDP HFA 80 µg/day; Placebo

SUMMARY:
This is a phase 2, randomized, double-blind, placebo-controlled, parallel-group, 2-week, multi-center, dose-range-finding study in male or female patients (12 years and older) with SAR.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients 12 years of age and older, as of the Screening Visit (SV).
* General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the study.
* A history of SAR to relevant seasonal allergen (tree/grass pollen) for a minimum of two years immediately preceding the study Screening Visit (SV). The SAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and in the investigator's judgment is expected to be exposed to the allergen and require treatment throughout the entire study period.
* A demonstrated sensitivity to relevant tree/grass pollen known to produce SAR through a standard skin prick test. A positive test is defined as a wheal diameter at least 3 mm larger than the control wheal for the skin prick test. Documentation of a positive result within 12 months prior to Screening Visit (SV) is acceptable.
* Other criteria apply

Key Exclusion Criteria:

* Participation in any investigational drug study within the 30 days preceding the Screening Visit (SV) or planned participation in another investigational drug study at any time during this study.
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma or surgery, atrophic rhinitis, or rhinitis medicamentosa (all within the last 60 days prior to the SV).
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, chronic sinusitis, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit (SV), or development of a respiratory infection during the Run-in Period.
* Use of any prohibited concomitant medications within the prescribed (per protocol) time since the last dosing period prior to the Screening Visit (SV) and/or plans for use during the entire treatment duration.
* Other criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, Ph.D., Study Chair — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (25):
- United States (25):
  - Teva Global Respiratory Research Study Site, Mission Viejo, California
  - Teva Global Respiratory Research Study Site, San Diego, California
  - Teva Global Respiratory Research Study Site, Colorado Springs, Colorado
  - Teva Global Respiratory Research Study Site, Denver, Colorado
  - Teva Global Respiratory Research Study Site, Gainesville, Georgia
  - Teva Global Respiratory Research Study Site, Savannah, Georgia
  - Teva Global Respiratory Research Study Site, Indianapolis, Indiana
  - Teva Global Respiratory Research Study Site, Overland Park, Kansas
  - Teva Global Respiratory Research Study Site, Bethesda, Maryland
  - Teva Global Respiratory Research Study Site, St Louis, Missouri
  - Teva Global Respiratory Research Study Site, Brick, New Jersey
  - Teva Global Respiratory Research Study Site, Raleigh, North Carolina
  - Teva Global Respiratory Research Study Site, Medford, Oregon
  - Teva Global Respiratory Research Study Site, Portland, Oregon
  - Teva Global Respiratory Research Study Site, Blue Bell, Pennsylvania
  - Teva Global Respiratory Research Study Site, Pittsburgh, Pennsylvania
  - Teva Global Respiratory Research Study Site, Upland, Pennsylvania
  - Teva Global Respiratory Research Study Site, Charleston, South Carolina
  - Teva Global Respiratory Research Study Site, Austin, Texas
  - Teva Global Respiratory Research Study Site, Dallas, Texas
  - Teva Global Respiratory Research Study Site, New Braunfels, Texas
  - Teva Global Respiratory Research Study Site, San Antonio, Texas
  - Teva Global Respiratory Research Study Site, Draper, Utah
  - Teva Global Respiratory Research Study Site, Burke, Virginia
  - Teva Global Respiratory Research Study Site, Richmond, Virginia

REFERENCES:
- [Derived] Raphael GD, Berger WE, Prenner BM, Finn AF Jr, Kelley L, Tantry SK. Efficacy, safety, and optimal dose selection of beclomethasone dipropionate nasal aerosol for seasonal allergic rhinitis in adolescents and adults. Curr Med Res Opin. 2013 Oct;29(10):1329-40. doi: 10.1185/03007995.2013.821055. Epub 2013 Aug 6. PMID 23815103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 685 patients were screened and 635 were enrolled in the study and participated in the Run-in Period. Of the 635 enrolled patients, 487 were randomized to treatment. The study was performed in the spring during tree and grass pollen seasons.
Pre-assignment Details: During the 7 - 21 day Run-in Period, patients self-administered a single-blind placebo nasal aerosol once daily in the morning and assessed and recorded their twice daily allergic rhinitis symptoms to determine eligibility for randomization.
Groups:
- BDP HFA 80 µg/Day: During the 2-week double-blind Treatment Period participants self-administered two actuations (one per nostril) of 40 micrograms (µg) beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) and two actuations of placebo HFA once daily.
Period: Overall Study
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Started | 118 | 123 | 122 | 124
Intent to Treat / Safety Population | 118 | 123 | 122 | 123 (One patient did not receive any double-blind study medication.)
Completed | 116 | 120 (One patient discontinued due to both an AE and study medication discontinuation.) | 120 | 114
Not Completed | 2 | 3 | 2 | 10
Not completed — Adverse Event | 0 | 1 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- BDP HFA 80 µg/Day: During the 2-week double-blind Treatment Period participants self-administered two actuations (one per nostril) of 40 (µg) BDP HFA and two actuations of placebo HFA once daily.
- Total: Total of all reporting groups
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo | Total
Number analyzed (Participants) | 118 | 123 | 122 | 123 | 486
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the Intent to Treat population.
  years | 37.6 (13.86) | 39.8 (15.26) | 38.5 (14.74) | 38.2 (13.95) | 38.5 (14.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 86 | 81 | 73 | 316
  Male | 42 | 37 | 41 | 50 | 170
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 92 | 99 | 98 | 97 | 386
  Black | 23 | 18 | 22 | 19 | 82
  Asian | 2 | 5 | 0 | 6 | 13
  Other | 1 | 1 | 2 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 10 | 17 | 15 | 56
  Not Hispanic or Latino | 104 | 113 | 105 | 108 | 430
Region of Enrollment [Number; unit: participants]
  United States | 118 | 123 | 122 | 123 | 486

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM and PM Reflective Total Nasal Symptom Score (rTNSS) Over the Two-week Treatment Period
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) over the past 12 hours twice daily (AM & PM) using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, easily tolerated); 2=moderate (awareness of sign/symptom, bothersome but tolerable); 3=severe (sign/symptoms hard to tolerate, interfere with daily activities and/or sleeping).
  The total nasal symptom score (sum of the 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Day -6 to 0) and Days 1-15 (2-week Treatment Period)
Population: The Intent-to-treat population included all randomized patients who received at least one dose of randomized study medication and had at least one post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 118 | 123 | 122 | 123
units on a scale | -1.88 (0.18) | -1.87 (0.18) | -2.22 (0.18) | -1.59 (0.18)
Statistical Analysis 1: Comparison: BDP HFA 80 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.255, Repeated measures ANCOVA — A multiplicity adjustment procedure was implemented which allowed for control of the Type I error within a particular treatment comparison, as well as within a particular endpoint, however it did not control the overall Type I error; The repeated measures ANCOVA included covariate adjustment for baseline, day, treatment, and the treatment by day interaction; LS Mean Difference = -0.29, 95% CI 2-sided [-0.80 to 0.21], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: BDP HFA 160 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.257, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.29, 95% CI 2-sided [-0.78 to 0.21], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: BDP HFA 320 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.013, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.63, 95% CI 2-sided [-1.13 to -0.13], Standard Error of Mean 0.25

2. Secondary Outcome: Change From Baseline in Average AM and PM Instantaneous Total Nasal Symptom Score (iTNSS) Over the Two Week Treatment Period
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) over the 10 minutes prior to the assessment, twice daily (AM & PM) using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, easily tolerated); 2=moderate (awareness of symptom, bothersome but tolerable); 3=severe (symptoms hard to tolerate, interfere with daily activities and/or sleeping). The total nasal symptom score (sum of 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Day -6 to 0) and Days 1-15 (2-week Treatment Period)
Population: Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 118 | 123 | 122 | 123
units on a scale | -1.77 (0.18) | -1.71 (0.18) | -2.10 (0.18) | -1.50 (0.18)
Statistical Analysis 1: Comparison: BDP HFA 80 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.278, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.77 to 0.22], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: BDP HFA 160 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.385, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.22, 95% CI 2-sided [-0.70 to 0.27], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: BDP HFA 320 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.016, Repeated Measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.60, 95% CI 2-sided [-1.09 to -0.11], Standard Error of Mean 0.25

3. Secondary Outcome: Change From Baseline in Morning Instantaneous Total Nasal Symptom Score (iTNSS) Over the Two-week Treatment Period
Description: Change from Baseline in the morning patient-reported instantaneous TNSS. Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) over the past 10 minutes (prior to the assessment) in the morning on a scale from 0 (mild symptoms) to 3 (severe symptoms). The total nasal symptom score (sum of the 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Day -6 to 0) and Days 1-15 (2-week Treatment Period)
Population: Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 118 | 123 | 122 | 123
units on a scale | -1.76 (0.18) | -1.71 (0.18) | -2.14 (0.18) | -1.31 (0.18)
Statistical Analysis 1: Comparison: BDP HFA 80 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.082, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.45, 95% CI 2-sided [-0.95 to 0.06], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: BDP HFA 160 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.114, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.90 to 0.10], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: BDP HFA 320 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.001, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.83, 95% CI 2-sided [-1.33 to -0.33], Standard Error of Mean 0.26

4. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: The adult RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional). Participants were asked to recall their experiences during the previous week and to give their responses on a 7-point scale (0 = Least severe to 6 = Extremely severe). The overall RQLQ score is the mean of all 28 responses, and ranges from 0 to 7. A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline and Week 2
Population: The RQLQ population included only those participants over the age of 18 years with an impaired quality of life at Baseline as defined by a RQLQ score at the Randomization Visit of 3.0 or greater.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 68 | 83 | 69 | 77
units on a scale | -1.30 (0.17) | -1.33 (0.15) | -1.62 (0.17) | -1.22 (0.16)
Statistical Analysis 1: Comparison: BDP HFA 80 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.747, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Results obtained from ANCOVA with treatment, baseline and center in the model; LS Mean Difference = -0.07, 95% CI 2-sided [-0.52 to 0.37], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: BDP HFA 160 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.605, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Results obtained from ANCOVA with treatment, baseline and center in the model; LS Mean Difference = -0.11, 95% CI 2-sided [-0.53 to 0.31], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: BDP HFA 320 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.083, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Results obtained from ANCOVA with treatment, baseline and center in the model; LS Mean Difference = -0.39, 95% CI 2-sided [-0.84 to 0.05], Standard Error of Mean 0.23

5. Secondary Outcome: Change From Baseline in Morning 24-hour Reflective Ocular Symptom Score Over the Two-week Treatment Period
Description: Participants recorded the severity of their symptoms (itching/burning eyes, tearing/watering eyes and redness of eyes) for the past 24 hours each morning using the following scale:
  0=absent (no sign/symptoms); 1=mild (sign/symptom present, minimal awareness, easily tolerated); 2=moderate (awareness of sign/symptom, bothersome but tolerable); 3=severe (sign/symptom hard to tolerate, interfere with daily activities or sleeping).
  The total ocular symptom score (sum of 3 symptom scores) ranges from 0 to 9 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Day -6 to 0) and Days 1-15 (2-week Treatment Period)
Population: The ocular population included only those participants with adequate ocular symptoms during the Run-in Period as defined by a mean daily 24-hour reflective score of 4 or greater for the 24-hour reflective ocular symptom score, over the last 7 days of the Run-in Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 95 | 102 | 101 | 100
units on a scale | -1.16 (0.16) | -1.11 (0.16) | -1.46 (0.16) | -1.17 (0.16)
Statistical Analysis 1: Comparison: BDP HFA 80 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.989, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.00, 95% CI 2-sided [-0.45 to 0.46], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: BDP HFA 160 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.808, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.06, 95% CI 2-sided [-0.39 to 0.50], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: BDP HFA 320 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.195, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.29, 95% CI 2-sided [-0.74 to 0.15], Standard Error of Mean 0.23

6. Secondary Outcome: Change From Baseline in Morning 24-hour Reflective Non-nasal Symptom Score Over the Two-week Treatment Period
Description: Participants recorded the severity of their symptoms (itching/burning eyes, tearing/watering eyes, redness of eyes and itching of ears or palate) for the past 24 hours each morning using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, easily tolerated); 2=moderate (awareness of sign/symptom, bothersome but tolerable); 3=severe (symptoms hard to tolerate, interfere with daily activities or sleeping).
  Total non-nasal symptom score (sum of 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from Baseline score indicates symptom improvement.
Time Frame: Baseline (Day -6 to 0) and Days 1-15 (2-week Treatment Period)
Population: The non-nasal population included only those participants with adequate non-nasal symptoms during the Run-in Period as defined by a mean daily 24-hour reflective score of 6 or greater for the 24-hour reflective non-nasal symptom score, over the last 7 days of the Run-in Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 92 | 94 | 97 | 97
units on a scale | -1.55 (0.22) | -1.49 (0.22) | -1.91 (0.21) | -1.51 (0.22)
Statistical Analysis 1: Comparison: BDP HFA 80 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.903, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.04, 95% CI 2-sided [-0.64 to 0.57], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: BDP HFA 160 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.952, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.02, 95% CI 2-sided [-0.58 to 0.62], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: BDP HFA 320 µg/Day vs Placebo; A priori threshold for statistical significance is p<0.05; Test type: Superiority or Other; p = 0.187, Repeated measures ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.99 to 0.19], Standard Error of Mean 0.30

ADVERSE EVENTS:
Arm/Group | BDP HFA 80 µg/Day | BDP HFA 160 µg/Day | BDP HFA 320 µg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/118 | 2/123 | 0/122 | 0/123
Other Adverse Events (participants affected / at risk) | 6/118 | 3/123 | 3/122 | 1/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 80 µg/Day (N=118) | BDP HFA 160 µg/Day (N=123) | BDP HFA 320 µg/Day (N=122) | Placebo (N=123)
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 80 µg/Day (N=118) | BDP HFA 160 µg/Day (N=123) | BDP HFA 320 µg/Day (N=122) | Placebo (N=123)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.